CLINICAL TRIAL: NCT03840174
Title: A Phase I Randomized, Double-Blind, Placebo-controlled Study to Evaluate the Safety, Tolerability and Immunogenicity of V160 (Human Cytomegalovirus Vaccine) in Healthy Japanese Men
Brief Title: Safety and Immunogenicity of the Human Cytomegalovirus (CMV) Vaccine (V160) in Healthy Japanese Men (V160-003)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: V160-003; V160-003 (Other: Merck Protocol Number); 194648 (Registry Identifier: JAPIC-CTI)
Record Dates: First submitted 2019-02-12; First posted 2019-02-15 (Actual); Results first posted 2021-11-15 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Cytomegalovirus Infections
MeSH Terms: conditions — Cytomegalovirus Infections

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- V160 (Experimental): Participants will receive V160 vaccination by IM injection on Day 1, Month 2, and Month 6.
  Interventions: Biological: V160
- Placebo (Placebo Comparator): Participants will receive placebo by IM injection on Day 1, Month 2, and Month 6.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: V160 — V160 administered as a 0.5 mL (100 Units) IM injection containing 225 mcg aluminum phosphate adjuvant (APA)
  Arms: V160
Other: Placebo — Saline solution (0.9% sodium chloride [NaCl] administered as a 0.5 mL IM injection
  Arms: Placebo

SUMMARY:
The purpose of the study is to assess the safety and tolerability of a 3-dose regimen of V160 administered by intramuscular (IM) injection in healthy Japanese male participants by cytomegalovirus (CMV) serostatus. There is no formal hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* Healthy based on medical history and physical examination
* Serologically confirmed to be CMV seropositive or CMV seronegative at Visit 1
* If of reproductive potential, agrees to the following from randomization through at least 4 weeks after the last dose of V160-/placebo (from Day 1 through Month 7): 1) practice abstinence from heterosexual activity and remain abstinent, or 2) use contraception unless confirmed to be azoospermic as detailed in the protocol

Exclusion Criteria:

* History of any allergic reaction or anaphylactic reaction to any vaccine component that required medical intervention
* Plans donation of sperm any time from signing the informed consent through 1 month after receiving the last dose of study drug
* Is currently immunocompromised or has been diagnosed as having a congenital or acquired immunodeficiency, human immunodeficiency virus (HIV) infection, lymphoma, leukemia, systemic lupus erythematosus, rheumatoid arthritis, juvenile rheumatoid arthritis, inflammatory bowel disease, or other autoimmune condition that requires immunosuppressive medication.
* Has a condition in which repeated venipuncture or injections post more than minimal risk for the participant, such as hemophilia, thrombocytopenia, other severe coagulation disorders, or significantly impaired venous access
* Has major psychiatric illness including: any history or schizophrenia or severe psychosis, bipolar disorder requiring therapy, or suicidal ideation within 3 years.
* Has previously received any CMV vaccine
* Had any live virus vaccine administered or scheduled to be administered in the period from 4 weeks prior to, and 4 weeks following receipt of study drug
* Had any inactivated vaccine administered or scheduled within the period from 14 days prior to, through 14 days following study drug
* Had administration of any immune globulin or blood product within 90 days prior to injection with study drug or scheduled within 30 days thereafter
* Has received systemic corticosteroids (equivalent of ≥2 mg/kg total daily dose of prednisone or ≥20 mg/d for persons weighing >10 kg) for ≥14 consecutive days and has not completed treatment at least 30 days prior to study entry
* Has received systemic corticosteroids exceeding physiologic replacement doses (≈5 mg/d prednisone equivalent) within 14 days prior to the first vaccination (participants using inhaled, nasal, or topical steroids are considered eligible for the study)
* Has received any anti-viral agent (e.g. letermovir, ganciclovir, valganciclovir, foscarnet, and valacyclovir) with proven or potential activity against CMV 14 days prior to vaccination or is likely to receive such an agent within 14 days after vaccination

  * Receiving or has received in the year prior to enrollment immunosuppressive therapies including but not limited to rapamycin (also sirolimus), tacrolimus (also FK-506), or other therapies used for solid organ/cell transplant, radiation therapy, immunosuppressive/cytotoxic immunotherapy, chemotherapy and other immunosuppressive therapies known to interfere with the immune response. Topical tacrolimus is allowed provided that it is not used within 14 days prior to, or 14 days following study drug
* Has participated in another clinical trial in the past 4 weeks, or plans to participate in a treatment-based trial or a trial in which an invasive procedure is to be performed while enrolled in this trial.

Ages: 20 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Healthy Japanese male participants between the ages of 20 and 64 (inclusive)
Enrollment: 18 (Actual)
Dates: Start 2019-03-08 (Actual); Primary Completion 2019-11-07 (Actual); Study Completion 2019-11-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- Souseikai PS Clinic ( Site 0001), Fukuoka, Japan

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Murata S, Oshima N, Iwasa T, Fukao Y, Sawata M. Safety, Tolerability, and Immunogenicity of V160, a Conditionally Replication-Defective Cytomegalovirus Vaccine, in Healthy Japanese Men in a Randomized, Controlled Phase 1 Study. Antibodies (Basel). 2023 Mar 10;12(1):22. doi: 10.3390/antib12010022. PMID 36975369

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy male participants 20 to 64 years of age were recruited at study sites in Japan.
Groups:
- V160: CMV Seronegative at Baseline: Participants who were cytomegalovirus (CMV)-seronegative at baseline received V160 vaccination by IM injection on Day 1, Month 2, and Month 6. V160 was administered as a 100-unit dose, with aluminum phosphate adjuvant.
- V160: CMV Seropositive at Baseline: Participants who were CMV-seropositive at baseline received V160 vaccination by IM injection on Day 1, Month 2, and Month 6. V160 was administered as a 100-unit dose, with aluminum phosphate adjuvant.
- Placebo: CMV Seronegative at Baseline: Participants who were CMV-seronegative at baseline received placebo by IM injection on Day 1, Month 2, and Month 6.
- Placebo: CMV Seropositive at Baseline: Participants who were CMV-seropositive at baseline received placebo by IM injection on Day 1, Month 2, and Month 6.
Period: Overall Study
Arm/Group | V160: CMV Seronegative at Baseline | V160: CMV Seropositive at Baseline | Placebo: CMV Seronegative at Baseline | Placebo: CMV Seropositive at Baseline
Started | 6 | 6 | 3 | 3
Vaccination 1 | 6 | 6 | 3 | 3
Vaccination 2 | 5 | 6 | 3 | 3
Vaccination 3 | 5 | 6 | 3 | 3
Completed | 5 | 6 | 3 | 3
Not Completed | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- V160: CMV Seronegative at Baseline: Participants who were CMV-seronegative at baseline received V160 vaccination by IM injection on Day 1, Month 2, and Month 6. V160 was administered as a 100-unit dose, with aluminum phosphate adjuvant.
- Total: Total of all reporting groups
Arm/Group | V160: CMV Seropositive at Baseline | Placebo: CMV Seropositive at Baseline | V160: CMV Seronegative at Baseline | Placebo: CMV Seronegative at Baseline | Total
Number analyzed (Participants) | 6 | 3 | 6 | 3 | 18
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.8 (16.4) | 36.3 (16.0) | 33.8 (11.5) | 24.7 (5.5) | 36.4 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 6 | 3 | 6 | 3 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 3 | 6 | 3 | 18
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 6 | 3 | 6 | 3 | 18
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Solicited Injection-site Adverse Event (AE)
Description: Participants used the vaccination report card (VRC) to document the presence of any solicited injection-site AEs (pain/tenderness, erythema/redness, and swelling) that occurred in the 5 days after each vaccination. The percentage of participants with a solicited injection-site AE was reported.
Time Frame: Up to 5 days after each vaccination
Population: All randomized participants who received at least 1 vaccination
Measure: Number; unit: Percentage of participants
Arm/Group | V160: CMV Seronegative at Baseline | V160: CMV Seropositive at Baseline | Placebo: CMV Seronegative at Baseline | Placebo: CMV Seropositive at Baseline
Number analyzed (Participants) | 6 | 6 | 3 | 3
Percentage of participants | 100.0 | 83.3 | 0.0 | 33.3

2. Primary Outcome: Percentage of Participants With a Solicited Systemic Adverse Event (AE)
Description: Participants used the vaccination report card (VRC) to document the presence of any solicited systemic AEs (headache, fatigue, muscle pain, joint pain) that occurred in the 14 days after each vaccination. The percentage of participants with a solicited systemic AE is reported.
Time Frame: Up to 14 days after each vaccination
Population: All randomized participants who received at least 1 vaccination
Measure: Number; unit: Percentage of participants
Arm/Group | V160: CMV Seronegative at Baseline | V160: CMV Seropositive at Baseline | Placebo: CMV Seronegative at Baseline | Placebo: CMV Seropositive at Baseline
Number analyzed (Participants) | 6 | 6 | 3 | 3
Percentage of participants | 33.3 | 16.7 | 33.3 | 66.7

3. Primary Outcome: Percentage of Participants With a Vaccine-related Serious Adverse Event (SAE)
Description: An SAE is defined as any untoward medical occurrence that, at any dose, results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; or other important medical event. The percentage of participants with an SAE considered to be at least possibly related to the study intervention will be reported
Time Frame: Up to 14 days after each vaccination
Population: All randomized participants who received at least 1 vaccination
Measure: Number; unit: Percentage of participants
Arm/Group | V160: CMV Seronegative at Baseline | V160: CMV Seropositive at Baseline | Placebo: CMV Seronegative at Baseline | Placebo: CMV Seropositive at Baseline
Number analyzed (Participants) | 6 | 6 | 3 | 3
Percentage of participants | 0.0 | 0.0 | 0.0 | 0.0

4. Secondary Outcome: Geometric Mean Titer (GMT) of CMV-specific Neutralizing Antibody (NAb)
Description: The NAb GMT in initially CMV-seronegative participants vaccinated with a 3-dose regimen of V160 administered IM was assessed.
Time Frame: 1 month after third vaccination (at 7 months)
Population: All randomized participants who were CMV-seronegative at baseline, received all 3 vaccinations, and did not deviate from the protocol in ways that could affect the immune response
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric Mean Titer
Arm/Group | V160: CMV Seronegative at Baseline | Placebo: CMV Seronegative at Baseline
Number analyzed (Participants) | 4 | 3
Geometric Mean Titer | 3651 [1688 to 7895] | NA [NA to 115] — Values below the lower limit of titer (<94) are represented by NA.
Statistical Analysis 1: Comparison: V160: CMV Seronegative at Baseline vs Placebo: CMV Seronegative at Baseline; Test type: Other; GMT Ratio = 77.7, 95% CI 2-sided [23.9 to 252.4] — Geometric Mean Titer (GMT) ratio and 95% CI were estimated using an ANOVA model

5. Secondary Outcome: Number of Participants With Viral Detection of V160 in Plasma
Description: The number of participants with positive viral detection in plasma (defined by viral load in plasma ≥assay defined threshold cutoff value) was assessed.
Time Frame: Day 1 (predose, at dosing, and 3 hours postdose), Day 3, Day 7, and Day 14
Population: All randomized participants who received at least one vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | V160: CMV Seronegative at Baseline | V160: CMV Seropositive at Baseline | Placebo: CMV Seronegative at Baseline | Placebo: CMV Seropositive at Baseline
Number analyzed (Participants) | 6 | 6 | 3 | 3
Participants
  Day 1 (predose) | 0 | 0 | 0 | 0
  0 min postdose in Day 1 | 1 | 0 | 0 | 0
  3 hr postdose in Day 1 | 0 | 0 | 0 | 0
  Day 3 postdose | 6 | 6 | 0 | 0
  Day 7 postdose | 0 | 0 | 0 | 0
  Day 14 postdose | 0 | 0 | 0 | 0

6. Secondary Outcome: Number of Participants With Wild-Type CMV Detection in Urine and Saliva
Description: The number of participants with positive wild-type viral shedding in urine or saliva (defined by viral load in saliva/urine ≥ assay defined threshold cutoff value) will be assessed.
Time Frame: Day 1 (predose), 3, 7, and 14 and Months 2, 6, and 7
Population: All randomized participants who received at least one vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | V160: CMV Seronegative at Baseline | V160: CMV Seropositive at Baseline | Placebo: CMV Seronegative at Baseline | Placebo: CMV Seropositive at Baseline
Number analyzed (Participants) | 6 | 6 | 3 | 3
Participants
  Day 1 (predose) | 0 | 0 | 0 | 0
  Day 3 (postdose [PD] 1) | 0 | 0 | 0 | 0
  Day 7 (PD1) | 0 | 0 | 0 | 0
  Day 14 (PD1) | 0 | 1 | 0 | 0
  Month 2 (predose 2) | 0 | 1 | 0 | 0
  Month 6 (predose 3) | 0 | 0 | 0 | 0
  Month 7 (PD3) | 0 | 1 | 0 | 0

7. Secondary Outcome: Number of Participants With Viral Detection of V160 in Injection-site Swab and Adhesive Tape Swab
Description: The number of participants with positive viral leakage in injection-site swab and adhesive tape swab (defined by viral load in injection-site swab/adhesive tape swab ≥ assay defined threshold cutoff value) will be assessed.
Time Frame: Day 1: 0, 10, 20, and 30 minutes postvaccination
Population: All randomized participants who received at least one vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | V160: CMV Seronegative at Baseline | V160: CMV Seropositive at Baseline | Placebo: CMV Seronegative at Baseline | Placebo: CMV Seropositive at Baseline
Number analyzed (Participants) | 6 | 6 | 3 | 3
Participants
  Swab from injection-site - 0 min PD1 | 6 | 6 | 0 | 0
  Swab from injection-site - 10 min PD1 | 3 | 4 | 0 | 0
  Swab from injection-site - 20 min PD1 | 4 | 4 | 0 | 0
  Swab from injection-site - 30 min PD1 | 3 | 4 | 0 | 0
  Swab from adhesive tape (inside) - 10 min PD1 | 1 | 2 | 0 | 0
  Swab from adhesive tape (inside) - 20 min PD1 | 0 | 3 | 0 | 0
  Swab from adhesive tape (inside) - 30 min PD1 | 0 | 0 | 0 | 0
  Swab from adhesive tape (outside) - 10 min PD1 | 0 | 0 | 0 | 0
  Swab from adhesive tape (outside) - 20 min PD1 | 0 | 0 | 0 | 0
  Swab from adhesive tape (outside) - 30 min PD1 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 14 days post each vaccination for AE/SAE, and up to 6.5 months for all-cause mortality.
Description: All randomized participants who received at least one vaccination are included in safety analysis.
Arm/Group | V160: CMV Seronegative at Baseline | V160: CMV Seropositive at Baseline | Placebo: CMV Seronegative at Baseline | Placebo: CMV Seropositive at Baseline
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 6/6 | 5/6 | 1/3 | 2/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V160: CMV Seronegative at Baseline (N=6) | V160: CMV Seropositive at Baseline (N=6) | Placebo: CMV Seronegative at Baseline (N=3) | Placebo: CMV Seropositive at Baseline (N=3)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (3) | 1 (1) | 1 (1) | 1 (1)
Injection site erythema (General disorders) | 3 (5) | 0 (0) | 0 (0) | 1 (1)
Injection site pain (General disorders) | 4 (10) | 5 (8) | 0 (0) | 1 (2)
Injection site swelling (General disorders) | 2 (3) | 1 (1) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-19): https://cdn.clinicaltrials.gov/large-docs/74/NCT03840174/Prot_SAP_000.pdf